CLINICAL TRIAL: NCT02612740
Title: Deproteinized Bovine Bone for the Treatment of Alveolar Bone Critical Size Defect in Humans: A Randomized Clinical Pilot Study
Brief Title: Deproteinized Bovine Bone in Alveolar Bone Critical Size Defect (>2cm) Secondary to Cyst Removal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Padova, School of Dental Medicine (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2187P
Record Dates: First submitted 2015-09-21; First posted 2015-11-24 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Maxillary Cyst
Keywords: Bio Oss; critical-size defect; bone grafting; cyst; CT bone analysis; alveolar bone
MeSH Terms: conditions — Cysts

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test Group (Experimental): The bone defect was filled with granules of deproteinized bovine bone (Bio-Oss, Geistlich Pharm, AG Wolhausen, Switzerland)
  Interventions: Biological: Deproteinized bovine bone; Device: granules of deproteinized bovine bone (Bio-Oss)
- Control Group (No Intervention): No filling material was used in the bone healing

INTERVENTIONS:
Biological: Deproteinized bovine bone — cyst removal followed by heterologous bone grafting
  Arms: Test Group
Device: granules of deproteinized bovine bone (Bio-Oss)
  Arms: Test Group

SUMMARY:
The aim of this study was to evaluate the effect of the use of deproteinized bovine bone as a filler material of critical-sized (diameter >=20 mm) bony defects derived from the excision of maxillary and mandibular cysts. 20 patients were considered.

Patients were randomly divided into 2 groups according to the type of treatment: the bone defect was filled with granules of deproteinized bovine bone (test); no filling material (control). Clinical parameters were recorded at 7 days, 1, 6 and 12 months after surgery. Radiological follow up consisted of an orthopantomograph and a CT scan taken at the baseline (pre-operatory) and 12 months after surgery.

In order to evaluate the difference in percentage of filling of the bone defect between the two groups, the pre-op and the 1-year radiolucent volumes were evaluated in the CT scans.

DETAILED DESCRIPTION:
The healing of extensive alveolar bone defects secondary to cyst removal is not predictable. Residual voids of various entity may persist. Some Authors proposed the use of grafting materials to reconstitute the loss of hard tissue. The primary objective was to determine the efficacy of bone grafting.The secondary objectives were to evaluate the incidence rate of wound dehiscence, pus drainage, recurrence and other complications 7 and 30 days and 6 months after surgery. Recurrence at 12 months of healing was also evaluated. For all patients included, surgeries were performed in conscious sedation and local anesthesia.Full-thickness flap of the appropriate shape and dimensions were lifted, and the bone exposed. When necessary, osteotomy was done, in order to enucleate the cystic lesion. The residual bone cavity was filled with deproteinized bovine bone (test), or not filled with any graft material (control). The flap was finally repositioned and sutured in order to achieve primary closure.

In both test and control groups antibiotic therapy with amoxicillin tablets of 1 g every 12 hours for six days (alternatively, for allergic patients, clarithromycin 500 mg tablets twice daily were given) and proper analgesics were prescribed. Postoperatory physical, therapy was prescribed as well.

Radiological follow up consisted of an orthopantomography and a CT scan taken at 12 months after surgery.For bone volume evaluation, a computerized method was adopted to compare the pre-operatory and the 12 months post-operatory CT scan. The Digital Imaging and Communication in Medicine (DICOM) obtained files were transferred to a Mac Pro Quad 2.66- GHz work- station (Apple Corp., Cupertino, CA, USA) and analyzed using an open-source medical image processing software (OsiriX v. 5.8.5, Pixmeo Sarl, Bernex, Switzerland). The margin of the radiolucent areas of each CT slice was traced manually on each axial view, and the volume calculated by the software with the ROI (Region Of Interest) tool. Volumes in mm3 and 3D images were obtained for each pre-op and post-op ct scan, for every test and control patient. Each exam was evaluated by two assessors (GL and SR) who were trained in radiological diagnosis and measurement detection. The volumetric reduction of the cysts was calculated by subtracting the preoperatory from the post operatory volumes, both in test and control groups.

ELIGIBILITY:
Inclusion Criteria:

* no smoking for at least 6 months;
* preoperative radiological diagnosis of radiolucent lesion of probable cystic origin;
* bone defect > 2 cm (diameter);
* ASA1;
* consent to the study inclusion.

Exclusion Criteria:

* subjects in need of treatment with a hemostatic material;
* active infection or inflammation in the treatment area;
* uncontrolled diabetes;
* bone diseases ( Paget's disease, patients undergoing bisphosphonate therapy, multiple myeloma, bone metastases);
* previous radiation therapy in the head and neck region;
* patients not able to take part to the follow-up program.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2014-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Bone volume evaluation | one year
  A computerized method was adopted to compare the pre-operatory and the 12 months post-operatory CT scan. The Digital Imaging and Communication in Medicine (DICOM) obtained files were transferred to a Mac Pro Quad 2.66- GHz work- station (Apple Corp., Cupertino, CA, USA) and analyzed using an open-source medical image processing software (OsiriX v. 5.8.5, Pixmeo Sarl, Bernex, Switzerland) (Lizio et al, 2013; Bittermann et al, 2014). The margin of the radiolucent areas of each CT slice was traced manually on each axial view, and the volume calculated by the software with the ROI (Region Of Interest) tool. Volumes in mm3 and 3D images were obtained for each pre-op and post-op ct scan, for every test and control patient. Each exam was evaluated by two assessors who were trained in radiological diagnosis and measurement detection. The volumetric reduction of the cysts was calculated by subtracting the preoperatory from the post operatory volumes, both in test and control groups.

SECONDARY OUTCOMES:
physiological parameter (wound dehiscence) | 7 days, 1, 6 and 12 months after surgery
  clinical evaluation (present/absent)
physiological parameter (pus drainage) | 7 days, 1, 6 and 12 months after surgery
  clinical evaluation (present/absent)
physiological parameter (recurrence) | 7 days, 1, 6 and 12 months after surgery
  clinical evaluation (present/absent)
physiological parameter (any other clinical complications) | 7 days, 1, 6 and 12 months after surgery
  clinical evaluation (present/absent)
bone density (scale - Hounsfield units) | 12 months after surgery
  Bone density analysis was conducted on three tomographic axial images (middle, caudal, cranial) of the healed cystic volume, per each patient of both groups. Bone density in Hounsfield Unit (HU) was obtained with the RadiAnt DICOM Viewer software (RadiAnt DICOM Viewer, version 1.1.8; Meixant, Poznan, Poland)